CLINICAL TRIAL: NCT02861898
Title: Phase I/II Trial of Super-selective Intra-arterial Repeated Infusion of Cetuximab for the Treatment of Newly Diagnosed Glioblastoma
Brief Title: Super-selective Intra-arterial Repeated Infusion of Cetuximab for the Treatment of Newly Diagnosed Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS16-0257
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma; Brain Cancer; Brain Neoplasm; Brain Tumor; Brain Neoplasm, Malignant; EGFR Gene Overexpression; GBM
Keywords: EGFR; Epidermal Growth Factor Receptor; EGFRvIII
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-arterial Cetuximab after BBBD (Experimental): Mannitol 20% 12.5ml over two minutes for Blood Brain Barrier (BBB) disruption followed by CTX administered intra-arterially for three doses at a dose of 250mg/m2
  Interventions: Drug: Intra-arterial Cetuximab; Drug: Intra-arterial Mannitol

INTERVENTIONS:
Drug: Intra-arterial Cetuximab
Drug: Intra-arterial Mannitol

SUMMARY:
Primary brain cancer kills up to 10,000 Americans a year. These brain tumors are typically treated by surgery, radiation therapy and chemotherapy, either individually or in combination. Present therapies are inadequate, as evidenced by the low 5-year survival rate for brain cancer patients, with median survival at approximately 12 months. Glioma is the most common form of primary brain cancer, afflicting approximately 7,000 patients in the United States each year. These highly malignant cancers remain a significant unmet clinical need in oncology. GBM often has a high expression EFGR (Epidermal Growth Factor Receptor) which is blocked by Cetuximab (CTX). The investigators have recently completed a separate Phase I clinical trial using superselective intra-arterial cerebral infusion (SIACI) of CTX after blood brain barrier disruption (BBBD) for recurrent GBM (Chakraborty et al, in revision, Journal of Neurooncology). The investigators found that intra-arterial infusion of CTX is well tolerated with few adverse effects. The investigators hypothesize that in patients with newly diagnosed GBM, repeated SIACI of this drug after BBBD will be safe and efficacious for our patients when combined with standard chemoradiation (STUPP protocol).

This trial will be a non-randomized open label Phase I/II clinical trial. In addition to standard chemotherapy and radiation therapy (STUPP protocol) the patient will be given CTX intra-arterially after BBBD for a total of three doses at approximately post surgery days 30, 120 and 210.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of ≥18 years of age.
* Patients with a documented histologic diagnosis of newly diagnosed glioblastoma multiforme (GBM)
* Patients with pathology confirmed histologic EGFR overexpression
* Patients must have at least one confirmed and evaluable tumor site.∗

  *A confirmed tumor site is one in which is biopsy-proven. NOTE: Radiographic procedures (e.g., Gd-enhanced MRI or CT scans) documenting existing lesions must have been performed within two weeks of treatment on this research study.
* Patients must have a Karnofsky performance status ≥70% (or the equivalent ECOG level of 0-2) and an expected survival of ≥ three months.
* No chemotherapy for two weeks prior to treatment under this research protocol and no external beam radiation for eight weeks prior to treatment under this research protocol.
* Patients must have adequate hematologic reserve with WBC≥3000/mm3, absolute neutrophils ≥1500/mm3 and platelets ≥100,000/ mm3. Patients who are on Coumadin must have a platelet count of ≥150,000/ mm3
* Pre-enrollment chemistry parameters must show: bilirubin<1.5X the institutional upper limit of normal (IUNL); AST or ALT<2.5X IUNL and creatinine<1.5X IUNL.
* Pre-enrollment coagulation parameters (PT and PTT) must be ≤1.5X the IUNL.
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study.
* Patients must be able to understand and give written informed consent. Informed consent must be obtained at the time of patient screening.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men will be informed as to the potential risk of conception while participating in this research trial and will be advised that they must use effective contraception during and for a period of three months after the treatment period.
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring
* Patients with radiological evidence of leptomeningeal disease.
* Patients with history of allergic reaction to CTX
* Patients who initiated or completed chemo/RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2016-06; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 6 months
  The 6-month PFS will be estimated by calculating the proportion of patients who are alive at 6 months from treatment commencement and are progression-free.
Overall Survival (OS) | 2 years
  OS will be calculated as the time from treatment initiation to the date of death.

SECONDARY OUTCOMES:
Composite overall response rate (CORR) through the Response Assessment in Neuro-Oncology (RANO) | 6 months
  Subjects will be classified according to the RANO criteria, which is a composite of MRI changes, clinical response and changes in steroid use.
Toxicities graded according to the NCI Common Toxicity Criteria (CTCAE) version 4.03 | 6 months
  Toxicities will be tabulated and graded according to the NCI Common Toxicity Criteria (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No